CLINICAL TRIAL: NCT00789360
Title: Pulmonary Safety of Repeat Doses of Staccato® Loxapine for Inhalation in Healthy Volunteers
Brief Title: Staccato Loxapine Pulmonary Safety in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMDC-004-104; 12 September 2008
Record Dates: First submitted 2008-11-07; First posted 2008-11-11 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2009-05

CONDITIONS: Healthy
Keywords: Healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inhaled Placebo crossed over to Inhaled Loxapine (Experimental): Inhaled Staccato Placebo, 2 inhalations, 8 hours apart; washout of at least 4 days; Inhaled Staccato Loxapine, 10 mg oses x 2, 8 hours apart
  Interventions: Drug: Inhaled Placebo; Drug: Inhaled Loxapine
- Inhaled Loxapine crossed over to Inhaled Placebo (Experimental): Inhaled Staccato Loxapine, 10 mg doses x 2, 8 hours apart; washout of at least 4 days; Inhaled Staccato Placebo, 2 inhalations, 8 hours apart;
  Interventions: Drug: Inhaled Placebo; Drug: Inhaled Loxapine

INTERVENTIONS:
Drug: Inhaled Placebo — Inhaled Staccato Placebo, 2 inhalations, 8 hours apart
Drug: Inhaled Loxapine — Inhaled Staccato Loxapine, 10 mg doses x 2, 8 hours apart

SUMMARY:
The objective of this trial is to assess the pulmonary safety of 2 inhaled doses of Staccato Loxapine within a day.

DETAILED DESCRIPTION:
The planned study is a multiple dose, double-blind, placebo-controlled, randomized, 2-sequence, 2-period crossover study investigating pulmonary safety in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* nonsmoker subjects in good general health with normal spirometry at screening AND baseline

Exclusion Criteria:

* history of asthma, COPD, or any other acute or chronic pulmonary disease or bronchodilator use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S. Miller, MD, Principal Investigator — Northeast Medical Research, North Dartmouth, MA
Locations (1):
- Northeast Medical Research, North Dartmouth, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Each investigator obtained approval from their IRB for their advertisements and other subject recruitment procedures
Pre-assignment Details: At screening and before administration of Dose 1 in each treatment period, the following were confirmed: forced expiratory volume in 1 second (FEV1) ≥85% of predicted, forced vital capacity (FVC) ≥85% of predicted, and oxygen saturation by pulse oximetry (SpO2)
  ≥95% on room air.
Groups:
- Inhaled Placebo / Loxapine: Inhaled Staccato Placebo, 2 inhalations, 8 hours apart followed by Inhaled Staccato Loxapine, 10 mg doses x 2, 8 hours apart
- Inhaled Loxapine / Placebo: Inhaled Staccato Loxapine, 10 mg oses x 2, 8 hours apart followed by Inhaled Staccato Placebo, 2 inhalations, 8 hours apart
Period: Overall Study
Arm/Group | Inhaled Placebo / Loxapine | Inhaled Loxapine / Placebo
Started | 15 | 15
Completed | 12 | 14
Not Completed | 3 | 1
Not completed — Protocol Violation | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Placebo / Loxapine | Inhaled Loxapine / Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (13.65) | 28.7 (9.75) | 30 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 10 | 10 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: The Largest Treatment Difference (Loxapine - Placebo) in Change in FEV1 From Baseline by Spirometry
Description: The largest treatment difference (Loxapine - Placebo) across the 17 post-treatment time points (15 min to 32 hr) in FEV1 Change from Same-Period Baseline,
Time Frame: 17 post-treatment time points (15 min to 32 hr)
Population: Crossover Spirometry Population (all subjects receiving both inhaled loxapine and inhaled placebo)
  LSM and CI statistics were based on the individual (within subject) differences between loxapine and placebo exposures
Measure: Least Squares Mean (90% Confidence Interval); unit: liters
Groups:
- Inhaled Staccato Placebo: Inhaled Staccato Placebo, 2 inhalations, 8 hours apart
Arm/Group | Inhaled Loxapine | Inhaled Staccato Placebo
Number analyzed (Participants) | 23 | 25
liters | -0.1042 [-0.1776 to -0.0310] | -0.1025 [-0.18099 to -0.02393]
Statistical Analysis 1: Comparison: Inhaled Loxapine vs Inhaled Staccato Placebo; The largest treatment difference (Loxapine - Placebo) in change in FEV1 from baseline by spirometry; Test type: Other; Maximum LS mean change difference = 0.0917, 90% CI 2-sided [-0.028 to 0.212] — Maximum difference occurred at 10 hours

2. Secondary Outcome: The Largest Treatment Difference (Loxapine - Placebo) in Change in FVC From Baseline by Spirometry
Description: The largest treatment difference (Loxapine - Placebo) across the 17 post-treatment time points (15 min to 32 hr) in FVC Change from Same-Period Baseline
Time Frame: 17 post-treatment time points (15 min to 32 hr)
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: liters
Groups:
- Inhaled Staccato: Inhaled Staccato Placebo, 2 inhalation, 8 hours apart
Arm/Group | Inhaled Loxapine | Inhaled Staccato
Number analyzed (Participants) | 25 | 25
liters | -0.271 [-0.370 to -0.172] | -0.149 [-0.264 to -0.035]
Statistical Analysis 1: Comparison: Inhaled Loxapine vs Inhaled Staccato; Test type: Other; Maximum LS mean change difference = -0.154, 90% CI 2-sided [-0.290 to -0.019] — Greatest difference occurred at 9 hours after Dose 1

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were considered treatment related from the first exposure to study treatment until 30 days after the last treatment
Description: Adverse events (AEs) were assessed predose and at 16 pre-specified time points for the 24-hour period after dosing, as well as whenever spontaneously reported by the subjects or study staff
Arm/Group | Inhaled Placebo | Inhaled Loxapine
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/29 | 0/27
Other Adverse Events (participants affected / at risk) | 5/29 | 16/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Placebo (N=29) | Inhaled Loxapine (N=27)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Placebo (N=29) | Inhaled Loxapine (N=27)
Dysgeusia (Gastrointestinal disorders) | 1 (1) | 12 (12)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less